CLINICAL TRIAL: NCT02574429
Title: Pilot Study Examining the Impact of a Cognitive Processing Therapy (CPT) Group for Patients With Co-Occurring Borderline Personality Disorder and Posttraumatic Stress Disorder
Brief Title: CPT Group for DBT Clients With Co-Occurring Borderline Personality Disorder and PTSD
Acronym: CPTDBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPTDBT-1
Record Dates: First submitted 2015-09-18; First posted 2015-10-12 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Borderline Personality Disorder; Posttraumatic Stress Disorder
Keywords: Borderline Personality Disorder; Posttraumatic Stress Disorder; Cognitive Processing Therapy; Group Therapy; Comorbidity; Dialectical Behavior Therapy
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Processing Therapy (Experimental): Individuals who have either completed Standard Dialectical Behavior Therapy (DBT) for Borderline Personality Disorder (BPD) and/or are currently enrolled in DBT who have co-occuring PTSD.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is an evidenced-based treatment for PTSD. The investigators are offering CPT group over 13 weeks (12 group sessions & 1 individual session). CPT focuses on challenging beliefs that developed or were reinforced following the trauma(s).
  Other Names: CPT

SUMMARY:
Even though borderline personality disorder (BPD) and posttraumatic stress disorder (PTSD) commonly co-occur, few studies have examined PTSD treatment among individuals with BPD. Additionally, many PTSD research studies exclude individuals with BPD due to their complexity and concerns regarding risk. This study aims to investigate the effectiveness of Cognitive-Processing Therapy Group (an evidenced-based treatment for PTSD) for individuals with these co-occurring disorders following completion of a Dialectical Behavioural Therapy Program (an evidenced-based treatment for BPD). The investigators are using a repeated measures pre and post design. Data will be collected prior to participants starting the CPT group, throughout the duration of the CPT group (i.e., weekly), and following the completion of the CPT group.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a severe psychological disorder characterized by instability in emotion regulation, interpersonal relationships, and self-image, coupled with marked impulsivity. Additionally, individuals with BPD often meet criteria for other disorders. One of the most commonly co-occurring disorders among individuals diagnosed with BPD is posttraumatic stress disorder (PTSD). Within this population, 56% to 58% of inpatients, and between 36% to 50% of outpatients are diagnosed with co-occurring PTSD.

The high prevalence of this co-occurrence is consistent with studies documenting the severe traumatic experiences (including, but not limited to, physical, sexual, and emotional abuse, both as children and adults) commonly experienced by individuals diagnosed with BPD . Additionally, risk factors for PTSD identified by meta-analyses share striking commonalities with those of BPD, including: lack of social support, prior history of trauma (including childhood abuse), and poor psychological adjustment prior to trauma.

The co-occurrence of BPD/PTSD is associated with poorer outcomes and significant distress than the presence of either disorder alone. For example, individuals with co-occurring BPD/PTSD exhibit a lower likelihood of remission from BPD after 10 years of follow-up, and are also more likely to engage in non-suicidal self-injurious behavior (NSSI). In addition, BPD patients diagnosed with PTSD are also faced with greater emotional dysfunction and global psychological distress, as well as inferior physical health compared to individuals with BPD alone.

Several studies have proposed theories on the high co-occurrence of these disorders, but few have investigated potential treatments to address the unique issues associated with this comorbidity. The current standard of treatment for BPD, Dialectical Behaviour Therapy (DBT), has a solid empirical basis, including numerous randomized control trials (RCTs) demonstrating its efficacy in the reduction of associated symptoms. Despite the efficacy of DBT, the DBT treatment manual (Linehan, 1993) did not outline a specific protocol for intervention in patients with co-occurring BPD and PTSD. Moreover, outcomes from DBT trials indicate that DBT alone does not adequately treat co-occurring BPD/PTSD. Specifically, data from an RCT evaluating DBT in suicidal women with BPD demonstrated that only 13% of patients diagnosed with BPD/PTSD achieved full remission from PTSD during one year of DBT.

Recently, researchers have focused on identifying how to treat individuals with BPD and PTSD within the context of DBT. Harned and colleagues have developed and tested a combined DBT PE protocol that has shown efficacy in treating BPD/PTSD. This combined treatment addresses some of the problems inherent in the direct application of the conventional PTSD treatment, prolonged exposure (PE) therapy for individuals with BPD. Evaluations of PE show that PE significantly reduces PTSD symptoms and secondary outcomes such as depression. PE is designed to counteract avoidance of traumatic memories through repeated exposure to the traumatic memory, as well as in vivo exposure to non-dangerous events perceived to be fearful by the patient. The intention of the treatment is to alleviate overestimation of the likelihood and severity of negative outcomes, as well as conditioned fear responses to certain situations, often experienced by PTSD patients.

Several characteristics of individuals with BPD interfere with the ability to engage in emotional exposure, the central intervention of PE therapy. These may include: self-injurious behaviours, other co-occurring issues (e.g. dissociation, substance use, ongoing trauma), emotional dysregulation (over-engagement, under-engagement, and strong non-fear emotions), trauma memory characteristics (large quantity and/or poor quality of trauma memories), and treatment noncompliance. The combined DBT protocol includes specific strategies to address these problems. While this combined DBT/PE protocol is an important step towards addressing the gap in treatment for individuals with co-occurring BPD/PTSD, there are other evidenced-based interventions that also merit evaluation in a combined DBT/PTSD treatment, notably Cognitive Processing Therapy (CPT).

Like PE, CPT has a strong evidence base to support its effectiveness treating PTSD. The protocol for CPT was initially generated as a treatment for victims of sexual assault and has since been successfully used to treat other types of trauma . It consists of cognitive therapy focused on how the traumatic event has impacted the individual's beliefs about themselves, others, and the world in general. The treatment involves 12 sessions of therapy, along with homework between sessions. The objective of the treatment is to first help patients identify dysfunctional beliefs and assumptions stemming from the traumatic experiences, challenge these beliefs (i.e., "stuck points", and then develop new beliefs reflecting a broader perspective.

While combined DBT/PE treatment is encouraging, CPT may have benefits that are similar to, if not superior to PE in some ways. Research on CPT indicates that treatment is similarly effective to PE in reducing PTSD symptoms and depression. However, their respective impact on secondary symptoms may differ due to the different mechanisms underlying each treatment. For example, one study suggested that CPT may be superior to PE on specific scales of guilt. One distinct benefit of CPT is that it is available and efficacious in both individual and group formats, whereas PE is available only individually. Group CPT allows efficient use of resources, which is critical in the context of a publicly funded health-system. In light of the fact that Standard DBT requires extensive clinician resources, the efficient use of supplementary treatments is even more critical. Finally, there may be other benefits to group that warrant research, including reduction of stigma of PTSD and associated shame by addressing this within a group context.

This study aims to assess the efficacy of CPT to address PTSD symptoms among individuals with co-occurring BPD/PTSD who are participating in Standard DBT. It is hypothesized that individuals will show significant reductions in primary symptom outcomes (PTSD) and secondary symptom outcomes (e.g., BPD symptoms, shame, anxiety, depression) between pre and post- treatment. This study aims to provide one of the first clinical examinations of the effectiveness of CPT as a treatment for co-occurring BPD and PTSD among individuals participating in Standard DBT. The results of such a trial could not only lead to the establishment a potentially clinically effective and cost-effective alternative to PE in this population, but also further elucidate the mechanism behind this complex comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with co-occurring BPD/PTSD who are either currently participating in Standard Dialectical Behaviour Therapy (DBT) or who have completed DBT

Exclusion Criteria:

-

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Weekly for 13 weeks (course of treatment)
  Self-report measure assessing change in PTSD DSM-5 symptoms are affecting the participant. The investigators are comparing pre-PCL scores to post-PCL scores. In addition, the investigators are interested in examing the pattern of change between sessions.

SECONDARY OUTCOMES:
BSL-23 | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-report measure assessing the presence of BPD symptoms (experiences and behaviors)
Ways of Coping Checklist (WCCL) | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-reported use of DBT skills use vs. less effective ways of coping
Depression, Anxiety, Stress and Suicide Scale (DASS-21) | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-report measure assessing symptoms of depression, anxiety, stress and suicide.
Difficulties in Emotion Regulation Scale (DERS) | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-report measure assessing how the individual expresses and copes with emotions
Experience of Shame Scale | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-report measure assessing the extent that an individual experienced shame
Anxiety Sensitivity Index (ASI-3) | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-report measure assessing the extent to which an individual is sensitive to anxiety cues
Self-compassion Scale (SCS) | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-report measure assessing the extent to which an individual treats his or herself self-compassionately.
The Life Events Checklist for DSM-5 (LEC-5) | Baseline only
  Self-reported description of the nature of the traumatic experience(s) the individual experienced.
Borderline Evaluation of Severity Overtime (BEST) | 2 times - once prior to starting treatment, and once at the end of 13 weeks of treatment
  Self-report measure assessing the presence of BPD symptoms (experiences and behaviors)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - St Joseph's Healthcare Hamilton, Community Psychiatry Clinic, Hamilton, Ontario